CLINICAL TRIAL: NCT01527149
Title: Ofatumumab (O) in Combination With Chemotherapy: Hyper-Fractionated Cyclophosphamide, Doxorubicin, Vincristine and Dexamethasone (O-HyperCVAD) Alternating With Ofatumumab High-Dose Cytarabine and Methotrexate (O-MA) for Patients With Newly Diagnosed Mantle Cell Lymphoma
Brief Title: Ofatumumab in Combination With Cyclophosphamide, Doxorubicin Hydrochloride, Vincristine Sulfate, and Dexamethasone Alternating With Ofatumumab in Combination With Cytarabine and Methotrexate in Treating Patients With Newly Diagnosed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 201611; NCI-2011-03562 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 201611 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2011-12-12; First posted 2012-02-06 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Stage I Mantle Cell Lymphoma; Stage II Contiguous Mantle Cell Lymphoma; Stage II Non-Contiguous Mantle Cell Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Methotrexate; merphos; ofatumumab; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (monoclonal antibody and combination chemotherapy) (Experimental): COURSES 1, 3, and 5 (O-HyperCVAD): Patients receive ofatumumab IV on day 1, cyclophosphamide IV over 2 hours every 12 hours for 6 doses on days 3-5, doxorubicin hydrochloride IV continuously over 72 hours on days 6-8, vincristine sulfate IV on days 6 and 13, and dexamethasone IV or PO on days 3-6 and 13-16.
  COURSES 2, 4, and 6 (O-HD-MA): Patients receive ofatumumab IV on day 1, methotrexate IV continuously over 24 hours on day 3, and cytarabine IV over 2 hours every 12 hours on days 4-5.
  All courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Eligible patients then undergo standard HDC-ASCT.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Biological: Ofatumumab; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous HDC-ASCT
  Other Names: Autologous Stem Cell Transplantation
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well ofatumumab in combination with cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and dexamethasone alternating with ofatumumab in combination with cytarabine and methotrexate works in treating patients with newly diagnosed mantle cell lymphoma (MCL). Monoclonal antibodies, such as ofatumumab, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, dexamethasone, cytarabine, and methotrexate, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ofatumumab together with alternating regimens of combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR), and in particular, the complete remission rate (CRR) in previously untreated MCL treated with ofatumumab in combination with aggressive chemo-immunotherapy.

SECONDARY OBJECTIVES:

I. To determine the high sensitivity flow cytometry (HSFCM) complete remission rate (HSFCM-CRR) in previously untreated MCL treated with ofatumumab in combination with aggressive chemo-immunotherapy +/- high dose chemotherapy and autologous stem cell transplant (HDC-ASCT).

II. To determine the time-to-progression (TTP), progression-free survival (PFS) and overall survival (OS) of patients with previously untreated MCL treated with ofatumumab and aggressive chemoimmunotherapy +/- HDC-ASCT.

III. To determine the toxicity profiles of ofatumumab in combination with high dose cytarabine chemoimmunotherapy +/- HDC-ASCT.

IV. To correlate minimal residual disease (MRD) at different time intervals with TTP, PFS, and OS.

V. To correlate surface cluster of differentiation (CD)20 levels, Ki67, and additional cytogenetic abnormalities in pretreatment tumor biopsies with respect to ORR, CRR, TTP, PFS, or OS.

VI. To determine the relationship between proliferation signature and clinical outcome using quantitative real-time reverse-transcriptase polymerase chain reaction (RT-PCR).

VII. To determine changes in surface CD20 levels, Ki67, or gain of additional cytogenetic abnormalities in relapsed/refractory tumor specimens.

VIII. To correlate serum component (C)3, C4, and hemolytic complement (CH)50 levels measured at baseline and at the end of first ofatumumab infusion with ORR, CRR, median response rate (MRR), TTP, PFS and OS.

IX. Evaluate the ability of the induction and consolidation therapy to get 70% of patients to autologous stem cell transplantation.

X. Evaluate the tolerability and CD34+ cell yield following therapy with patient and hyper-fractionated cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and dexamethasone (HyperCVAD)/high-dose cytarabine and methotrexate (HD-MA).

XI. To compare differences in response rate in patients with MCL treated with ofatumumab + HyperCVAD/HD-MA according Cheson and Modified Cheson Criteria.

OUTLINE:

COURSES 1, 3, and 5 (O-HyperCVAD): Patients receive ofatumumab intravenously (IV) on day 1, cyclophosphamide IV over 2 hours every 12 hours for 6 doses on days 3-5, doxorubicin hydrochloride IV continuously over 72 hours on days 6-8, vincristine sulfate IV on days 6 and 13, and dexamethasone IV or orally (PO) on days 3-6 and 13-16.

COURSES 2, 4, and 6 (O-HD-MA): Patients receive ofatumumab IV on day 1, methotrexate IV continuously over 24 hours on day 3, and cytarabine IV over 2 hours every 12 hours on days 4-5.

Treatment repeats every 21 days for 6* courses in the absence of disease progression or unacceptable toxicity.

Eligible patients then undergo standard high dose chemotherapy and autologous stem cell transplant (HDC-ASCT). Patients achieving a high sensitivity flow cytometry complete remission (HSFCM-CR) after 2 courses may proceed to HDC-ASCT after completing 4 courses of treatment.

After completion of study treatment, patients are followed up every 4 months for 2 years, every 6 months for 3 years, and then as clinically instructed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented mantle cell lymphoma with co-expression of CD20 and CD5 and lack of CD23 expression by immunophenotyping and at least one of the following confirmatory tests: 1) positive immunostaining for cyclin D1; 2) the presence of t(11;14) on cytogenetic analysis; OR 3) molecular evidence of B-cell leukemia/lymphoma 1 (bcl-1)/immunoglobulin heavy locus (IgH) rearrangement

  * Cases that are CD5-negative and/or CD23-positive will be eligible provided that the histopathology is consistent with mantle cell lymphoma AND positive for cyclin D1, t(11;14), or bcl-1/IgH rearrangement
  * A tissue block or unstained slides (10 - 20 slides) will be submitted to the Roswell Park Cancer Institute (RPCI) Pathology Department for central pathology review
  * A diagnosis based on peripheral blood or bone marrow aspirate is allowed; if the diagnosis is based only on blood, in addition to the immunophenotype and molecular confirmation above, a peripheral blood smear must be available for central pathology review; if the diagnosis is based on a bone marrow, the bone marrow core biopsy or aspirate clot tissue block will be submitted to the RPCI Pathology Department: if the tissue block is not available please submit the diagnostic smears for review
* Extent of disease: stage I - IV; patients with nodular histology mantle cell lymphoma must have Ann Arbor stage III or IV disease to be eligible

  * Patients with mantle zone type histology will not be eligible
  * Patients with other mantle cell histologies are eligible regardless of stage
* Measurable or assessable disease is required; measurable tumor size (at least one node measuring 2.25 cm^2 in bidimensional measurement)
* No active central nervous system (CNS) disease defined as symptomatic meningeal lymphoma or known CNS parenchymal lymphoma; a lumbar puncture demonstrating mantle cell lymphoma at the time of registration to this study is not an exclusion for study enrollment
* Patients must be previously untreated
* No prior radiation therapy for mantle cell lymphoma
* >= 2 weeks since major surgery
* No known hypersensitivity to murine products
* No medical condition requiring chronic use of high dose systemic corticosteroids (i.e., doses of prednisone higher than 10 mg/day or equivalent)
* No human immunodeficiency virus (HIV) infection; patients with a history of intravenous drug abuse or any behavior associated with an increased risk of HIV infection should be tested for exposure to the HIV virus; patients who test positive or who are known to be infected are not eligible; an HIV test is not required for entry on this protocol, but is required if the patient is perceived to be at risk
* Non-pregnant and non-nursing; women and men of reproductive potential should agree to use an effective means of birth control
* Patients who test positive for hepatitis C antibody (Ab) are eligible provided all of the following criteria are met: 1) total bilirubin =< 2 x upper limit of normal; 2) AND aspartate aminotransferase (AST) =< 3 x upper limit of normal; AND 3) liver biopsy (pathology) demonstrates =< grade 2 fibrosis and no cirrhosis
* Specific guidelines will be followed regarding inclusion of MCL based on hepatitis B serological testing as follows:

  * Hepatitis B surface antigen (HBsAg) negative, hepatitis B core antibody (HBcAb) negative, hepatitis B surface antibody (HBsAb) positive MCL patients are eligible
  * Patients who test positive for HBsAg are ineligible (regardless of other hepatitis B serologies)
  * For MCL patients with HBsAg negative, but HBcAb positive (regardless of HBsAb status), should have hepatitis B virus (HBV) deoxyribonucleic acid (DNA) testing done and protocol eligibility determined as follows:

    * If HBV DNA is positive the subject is excluded
    * If HBV DNA is negative, patient may be included but must undergo at least every 2 months HBV DNA polymerase chain reaction (PCR) testing from the start of treatment throughout the duration the study
    * Monitoring during the study is required at least every 2 months and during follow-up at a minimum of every 2-3 months up to 6 months after the last dose
    * Prophylactic antiviral therapy with lamivudine (3TC) or investigator's preferred antiviral regimen throughout protocol therapy and for 6-12 months thereafter may be initiated at the discretion of the investigator
    * If the patients' HBV DNA becomes positive during the study, the investigator should manage the clinical situation as per the standard of care of participating institution; the investigator should weigh the risks and benefits of continuing ofatumumab or discontinuing ofatumumab before appropriate treatment decisions are made for that individual patient
* Patients must not have a history of cardiac disease, defined as New York Heart Association class II or greater or clinical evidence of congestive heart failure (CHF)
* No known hypersensitivity to ofatumumab, humanized antibodies or chemotherapy agents throughout the protocol
* Left ventricular ejection fraction (LVEF) by multi gated acquisition scan (MUGA) or echocardiogram (ECHO) >= 45%
* Neutrophils > 1000/uL
* Platelets >= 75,000/uL (unless significant bone marrow involvement with MCL)
* Creatinine =< 2.0 mg/dL
* Total bilirubin =< 2.0 mg/dL (unless MCL related or attributable to Gilbert's disease)
* Urine or serum beta-human chorionic gonadotropin (HCG) or serum HCG = negative (if female patient of childbearing potential)
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Consult with a physician experience in care and management of subjects with hepatitis B to manage/treat subjects who are anti-hepatitis B core antibody (HBc) positive

Exclusion Criteria:

* Prior history of HIV-positivity (routine HIV testing is not required pre-treatment)
* Positive serology for hepatitis B (HB) defined as a positive test for HBsAg; in addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a hepatitis B DNA test will be performed and if positive the patient will be excluded
* Serious non-malignant disease (e.g., active uncontrolled bacterial, viral, or fungal infections) or other medical conditions (including psychiatric) which, in the opinion of the Principal Investigator (PI) would compromise other protocol objectives
* Presence of symptomatic CNS lymphoma
* Pregnant or lactating females
* Prior history of radiation or chemotherapy for MCL
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ofatumumab or other agents used in study
* Patients with a "currently active" second malignancy, other than non-melanoma skin cancer or in situ carcinoma of the cervix or breast; patients are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy, are considered by their physician to be at less than 30% risk of relapse and at least 2-5 years have lapsed
* Major surgery, other than diagnostic surgery, within 2 weeks
* Patients with non-Hodgkin lymphoma (NHL) other than MCL
* Patients must not have a history of cardiac disease, defined as New York Heart Association class II or greater or clinical evidence of congestive heart failure; all patients must have a MUGA scan or 2-dimensional (D) echocardiogram indicating an ejection fraction of >= 45% within 42 days prior to registration; the method used at baseline must be used for later monitoring
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-12-06 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2024-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Hernandez-ILizaliturri, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Torka P, Akhtar OS, Reddy NM, Baysal BE, Kader A, Groman A, Nichols J, Mavis C, Tario JD, Block AW, Sait SNJ, Ghione P, Sundaram S, Przespolewski ER, Mohr A, Lund I, Kostrewa J, McWhite K, DeMarco J, Johnson M, Darrall A, Thomas-Talley RN, Wallace PK, Neppalli V, Hutson A, Hernandez-Ilizaliturri FJ. Ofatumumab plus HyperCVAD/HD-MA induction leads to high rates of minimal residual disease negativity in patients with newly diagnosed mantle cell lymphoma: Results of a phase 2 study. Cancer. 2022 Apr 15;128(8):1595-1604. doi: 10.1002/cncr.34106. Epub 2022 Feb 14. PMID 35157306
- [Derived] Barth MJ, Mavis C, Czuczman MS, Hernandez-Ilizaliturri FJ. Ofatumumab Exhibits Enhanced In Vitro and In Vivo Activity Compared to Rituximab in Preclinical Models of Mantle Cell Lymphoma. Clin Cancer Res. 2015 Oct 1;21(19):4391-7. doi: 10.1158/1078-0432.CCR-15-0056. Epub 2015 May 11. PMID 25964296

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Monoclonal Antibody and Combination Chemotherapy): COURSES 1, 3, and 5 (O-HyperCVAD): Patients receive ofatumumab IV on day 1, cyclophosphamide IV over 2 hours every 12 hours for 6 doses on days 3-5, doxorubicin hydrochloride IV continuously over 72 hours on days 6-8, vincristine sulfate IV on days 6 and 13, and dexamethasone IV or PO on days 3-6 and 13-16.
  COURSES 2, 4, and 6 (O-HD-MA): Patients receive ofatumumab IV on day 1, methotrexate IV continuously over 24 hours on day 3, and cytarabine IV over 2 hours every 12 hours on days 4-5.
  All courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Eligible patients then undergo standard HDC-ASCT.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous HDC-ASCT
  Cyclophosphamide: Given IV
  Cytarabine: Given IV
  Dexamethasone: Given IV or PO
  Doxorubicin Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Methotrexate: Given IV
  Ofatumumab: Given IV
  Vincristine Sulfate: Given IV
Period: Overall Study
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Started | 37
Completed | 35
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Experiencing a Complete Response
Description: Evaluated according to the International Working Group Response criteria as reported by Cheson et al. and the revised Cheson criteria.
  Complete response is defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. Typically FDG-avid lymphoma: in patients with PET scan positive before therapy, a posttreatment residual mass of any size is permitted as long as it is PET negative. Variably FDG-avid lymphomas/FDG avidity unknown: in patients with a negative pretreatment PET scan, all lymph nodes and nodal masses must have regressed on CT to normal size (1.5 cm in their greatest transverse diameter for nodes 1.5 cm before therapy). Previously involved nodes that were 1.1 cm to 1.5 cm in their long axis and more than 1)
Time Frame: 22 weeks
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 37
Proportion of participants | .62 [.45 to .78]

2. Secondary Outcome: Percentage of Participants With Autologous Stem Cell Transplantation
Description: Estimated using simple relative frequencies. The corresponding 95% confidence intervals will be computed using the method proposed in Clopper and Pearson.
Time Frame: Up to 6 weeks after the last dose of ofatumumab-chemotherapy, an average of 4 month
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 37
percentage of participants | 73 [55 to 86]

3. Secondary Outcome: Change From Baseline in Percentage of Cells Positive for Ki67
Description: Mean change from baseline in Percentage of Cells Positive for Ki67 by patient response.
Time Frame: Baseline and up to 3 years
Population: All treated and eligible patients that had samples taken after baseline
Measure: Mean (Standard Deviation); unit: percentage of cells positive for Ki-67
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 2
percentage of cells positive for Ki-67
  Not CR | -2.5 (10.6)
  CR | NA (NA) — No patients with Ki67 measures after baseline had CR

4. Secondary Outcome: Median of Serum Complement CD20 Levels
Description: Median serum C20 MFI (mean fluorescence intensity)
Time Frame: Baseline
Population: All treated and evaluable patients
Measure: Median (Full Range); unit: mean fluorescence intensity
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 19
mean fluorescence intensity | 186.8 [0.0 to 480.2]

5. Secondary Outcome: Number of Participants With at Least One Serious Adverse Event
Description: Evaluated using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 3 years
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 37
Participants | 19

6. Secondary Outcome: Minimal Residual Disease (MRD) in Peripheral Blood Samples
Description: Minimal residual disease (MRD) in peripheral blood samples at baseline.
Time Frame: Up to 3 years
Population: All treated and eligible patients with available samples
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 31
Participants
  Negative | 2
  Postive | 29

7. Secondary Outcome: Minimal Residual Disease (MRD) in Bone Marrow Biopsy/Aspiration Samples
Description: Minimal residual disease (MRD) in and bone marrow biopsy/aspiration samples at baseline.
Time Frame: Up to 3 years
Population: All treated and eligible patients with available samples
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 30
Participants
  Negative | 6
  Postive | 24

8. Secondary Outcome: Median Overall Survival (OS)
Description: Estimated distributions obtained using the Kaplan-Meier method. Estimates of quantities such as median survival will be obtained. Corresponding confidence intervals using the methodology of Brookmeyer and Crowley will be computed.
Time Frame: From baseline through study completion, an average of 5 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 37
months | 56.0 [39.8 to 78.0]

9. Secondary Outcome: Median Progression-free Survival (PFS)
Description: as for outcome 8
Time Frame: From baseline through study completion, an average of 5 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 37
months | 45.5 [21.4 to 78.0]

10. Secondary Outcome: Proliferation Signature Using Quantitative Real-time RT-PCR
Description: Relationship between proliferation signature and clinical outcome will be compared using the log-rank test. Cox proportional hazards model regression will be utilized for multivariate analyses.
Time Frame: Baseline
Population: Samples were not viable due to inadequate tissue.
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 0

11. Secondary Outcome: Proportion of Patients Who Experience Complete Remission as Assessed by HSFCM
Description: Established when all CR criteria are met and negative flow cytometry examination of peripheral blood and bone marrow biopsy/aspiration collected at baseline, before courses 3 and 5, within 3 weeks after course 6, on day 100 (if HDC-ASCT eligible), and then every 6 months for 3 years.
Time Frame: Up to 3 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 37
Proportion of participants | .84 [.68 to .94]

12. Secondary Outcome: Time-to-tumor Progression (TTP) at 3 Years
Description: Estimated percentage of patients that progressed at 3 years. Time to Progression distributions obtained using the Kaplan-Meier method. Corresponding confidence intervals using the methodology of Brookmeyer and Crowley will be computed.
Time Frame: From baseline until objective tumor progression, as assessed up to 3 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
Number analyzed (Participants) | 37
percentage of participants | 76 [57 to 87]

ADVERSE EVENTS:
Time Frame: From the start date of intervention through study completion, an average of 5 years
Arm/Group | Treatment (Monoclonal Antibody and Combination Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 16/37
Serious Adverse Events (participants affected / at risk) | 19/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody and Combination Chemotherapy) (N=37)
Acute coronary syndrome (Cardiac disorders) | 1 (6)
Periorbital oedema (Eye disorders) | 1 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (4)
Pyrexia (General disorders) | 1 (6)
Diverticulitis (Infections and infestations) | 1 (6)
Enterocolitis infectious (Infections and infestations) | 1 (6)
Infusion site infection (Infections and infestations) | 3 (17)
Lung infection (Infections and infestations) | 2 (12)
Neutropenic sepsis (Infections and infestations) | 1 (3)
Parainfluenzae virus infection (Infections and infestations) | 1 (6)
Pneumonia (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 8 (56)
Neutrophil count decreased (Investigations) | 1 (6)
Cytarabine syndrome (Musculoskeletal and connective tissue disorders) | 1 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (12)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4)
Arachnoiditis (Nervous system disorders) | 1 (6)
Headache (Nervous system disorders) | 1 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Blister (Skin and subcutaneous tissue disorders) | 1 (6)
Hypotension (Vascular disorders) | 1 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody and Combination Chemotherapy) (N=37)
Anaemia (Blood and lymphatic system disorders) | 31 (291)
Febrile neutropenia (Blood and lymphatic system disorders) | 15 (51)
Leukopenia (Blood and lymphatic system disorders) | 2 (9)
Lymph node pain (Blood and lymphatic system disorders) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (37)
Atrial fibrillation (Cardiac disorders) | 2 (6)
Cardiac failure congestive (Cardiac disorders) | 1 (2)
Pericarditis (Cardiac disorders) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (2)
Tachycardia (Cardiac disorders) | 3 (8)
External ear inflammation (Ear and labyrinth disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (3)
Dry eye (Eye disorders) | 4 (10)
Eye disorder (Eye disorders) | 1 (3)
Eye haemorrhage (Eye disorders) | 1 (3)
Eye pain (Eye disorders) | 1 (2)
Lacrimation increased (Eye disorders) | 2 (6)
Periorbital oedema (Eye disorders) | 4 (12)
Photophobia (Eye disorders) | 1 (2)
Vision blurred (Eye disorders) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (5)
Abdominal pain (Gastrointestinal disorders) | 5 (19)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2)
Anal haemorrhage (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 18 (46)
Diarrhoea (Gastrointestinal disorders) | 10 (42)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 8 (23)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 4 (10)
Gastritis (Gastrointestinal disorders) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (15)
Lip dry (Gastrointestinal disorders) | 2 (5)
Nausea (Gastrointestinal disorders) | 28 (128)
Oesophagitis (Gastrointestinal disorders) | 1 (2)
Oral disorder (Gastrointestinal disorders) | 1 (2)
Proctalgia (Gastrointestinal disorders) | 1 (3)
Stomatitis (Gastrointestinal disorders) | 9 (44)
Vomiting (Gastrointestinal disorders) | 17 (73)
Adverse drug reaction (General disorders) | 1 (2)
Asthenia (General disorders) | 2 (5)
Catheter site oedema (General disorders) | 1 (3)
Catheter site pain (General disorders) | 1 (2)
Chest pain (General disorders) | 4 (11)
Chills (General disorders) | 3 (7)
Face oedema (General disorders) | 1 (2)
Fatigue (General disorders) | 15 (48)
Influenza like illness (General disorders) | 1 (4)
Infusion site erythema (General disorders) | 1 (3)
Infusion site haemorrhage (General disorders) | 1 (3)
Infusion site pain (General disorders) | 1 (2)
Infusion site rash (General disorders) | 2 (4)
Infusion site reaction (General disorders) | 1 (2)
Injection site reaction (General disorders) | 1 (3)
Localised oedema (General disorders) | 4 (13)
Malaise (General disorders) | 1 (3)
Mucosal inflammation (General disorders) | 2 (6)
Non-cardiac chest pain (General disorders) | 1 (2)
Oedema (General disorders) | 2 (4)
Oedema peripheral (General disorders) | 15 (38)
Pain (General disorders) | 8 (18)
Pyrexia (General disorders) | 17 (106)
Cytokine release syndrome (Immune system disorders) | 1 (4)
Hypersensitivity (Immune system disorders) | 2 (4)
Anorectal infection (Infections and infestations) | 1 (3)
Cellulitis (Infections and infestations) | 1 (3)
Diverticulitis (Infections and infestations) | 1 (3)
Influenza (Infections and infestations) | 1 (3)
Lung infection (Infections and infestations) | 1 (2)
Pharyngitis (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 1 (3)
Pseudomonas infection (Infections and infestations) | 1 (3)
Septic embolus (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (3)
Skin infection (Infections and infestations) | 1 (3)
Tuberculosis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (12)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 29 (87)
Skin laceration (Injury, poisoning and procedural complications) | 1 (3)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (4)
Activated partial thromboplastin time prolonged (Investigations) | 1 (3)
Alanine aminotransferase increased (Investigations) | 7 (17)
Aspartate aminotransferase increased (Investigations) | 6 (16)
Blood bilirubin increased (Investigations) | 3 (22)
Blood creatinine increased (Investigations) | 4 (44)
Blood magnesium decreased (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 2 (29)
Neutrophil count decreased (Investigations) | 16 (196)
Platelet count decreased (Investigations) | 32 (345)
Weight decreased (Investigations) | 4 (13)
White blood cell count decreased (Investigations) | 9 (104)
Decreased appetite (Metabolism and nutrition disorders) | 9 (23)
Dehydration (Metabolism and nutrition disorders) | 1 (3)
Fluid overload (Metabolism and nutrition disorders) | 12 (54)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 4 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (41)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (4)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (18)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 17 (143)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (21)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (11)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (4)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (29)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Cytarabine syndrome (Musculoskeletal and connective tissue disorders) | 1 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (9)
Dizziness (Nervous system disorders) | 5 (16)
Dysgeusia (Nervous system disorders) | 11 (30)
Dysmetria (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 17 (68)
Lethargy (Nervous system disorders) | 1 (3)
Neuropathy peripheral (Nervous system disorders) | 2 (5)
Paraesthesia (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (12)
Syncope (Nervous system disorders) | 1 (3)
Taste disorder (Nervous system disorders) | 1 (2)
Tremor (Nervous system disorders) | 1 (2)
Thrombosis in device (Product Issues) | 1 (3)
Anxiety (Psychiatric disorders) | 10 (26)
Confusional state (Psychiatric disorders) | 2 (5)
Depression (Psychiatric disorders) | 4 (9)
Insomnia (Psychiatric disorders) | 7 (18)
Acute kidney injury (Renal and urinary disorders) | 1 (13)
Dysuria (Renal and urinary disorders) | 2 (5)
Haematuria (Renal and urinary disorders) | 1 (3)
Pollakiuria (Renal and urinary disorders) | 2 (5)
Urinary retention (Renal and urinary disorders) | 3 (9)
Urinary tract pain (Renal and urinary disorders) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (20)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (38)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (8)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (10)
Blister (Skin and subcutaneous tissue disorders) | 1 (3)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (15)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (14)
Rash (Skin and subcutaneous tissue disorders) | 3 (12)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (20)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (11)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (6)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 2 (6)
Embolism (Vascular disorders) | 1 (2)
Flushing (Vascular disorders) | 1 (3)
Hypertension (Vascular disorders) | 3 (7)
Hypotension (Vascular disorders) | 5 (13)
Jugular vein thrombosis (Vascular disorders) | 2 (6)

LIMITATIONS AND CAVEATS:
Samples were not viable for some of the outcomes the due to inadequate tissue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT01527149/Prot_SAP_000.pdf